CLINICAL TRIAL: NCT01108341
Title: An Open-Label Study to Evaluate the Efficacy and Safety of Treatment With Bendamustine in Combination With Ofatumumab in Previously Untreated Patients With Indolent B-Cell Non-Hodgkin's Lymphoma (NHL)
Brief Title: Study to Evaluate the Efficacy and Safety of Treatment With Bendamustine in Combination With Ofatumumab in Previously Untreated Patients With Indolent B-Cell Non-Hodgkin's Lymphoma (NHL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C18083/2048; 2009-016725-34 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-22 (Estimated); Results first posted 2012-08-28 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-07

CONDITIONS: Non-Hodgkin's Lymphoma (NHL)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bendamustine and Ofatumumab (Experimental): There are 6 planned and 2 optional 28-day cycles in which participants are administered both bendamustine and ofatumumab in the following doses: Bendamustine administered at 90 mg/m^2 intravenously (iv) on study days 1 and 2. Ofatumumab administered at 300 mg iv on day 1 and 1000 mg iv on day 8 of cycle 1. Ofatumumab administered at 1000 mg iv on day 1 of all additional cycles.
  Interventions: Drug: Bendamustine hydrochloride; Drug: Ofatumumab

INTERVENTIONS:
Drug: Bendamustine hydrochloride — Bendamustine will be administered at 90 mg/m^2 as a 30-minute intravenous (iv) infusion on days 1 and 2 of each cycle.
  Other Names: CEP-18083; Treanda
Drug: Ofatumumab — Ofatumumab will be administered at 300 mg as an iv infusion on day 1 and 1000 mg on day 8 of cycle 1 and 1000 mg on day 1 of each subsequent cycle.
  Other Names: Arzerra

SUMMARY:
The primary objective of the study is to determine the efficacy, as measured by overall response (complete response + partial response) of bendamustine in combination with ofatumumab in previously untreated patients with indolent B-Cell Non-Hodgkin's Lymphoma (NHL).

ELIGIBILITY:
Key Inclusion Criteria:

* The patient has histopathologic confirmation of one of the protocol-specific CD20+ B-cell non-Hodgkin's lymphomas. Tissue diagnostic procedures must be performed within 6 months of study entry and with biopsy material available for review.
* The patient meets 1 of the following need-for-treatment criteria:

  1. Presence of at least 1 of the following B-symptoms:

     * fever (>38ºC) of unclear etiology
     * night sweats
     * weight loss of greater than 10% within the prior 6 months
  2. large tumor mass (bulky disease) characterized by lymphomas with a diameter of more than 3 cm in 3 or more regions or by a lymphoma with a diameter of more than 7 cm in 1 region
  3. presence of lymphoma-related complications
  4. hyperviscosity syndrome due to monoclonal gammopathy
* The patient's tumor is verified to be CD20+ positive from current or previous excisional or incisional tissue diagnostic procedures performed within 6 months of study entry.
* The screening phase CT scan (based on local evaluation) shows:
* 2 or more clearly demarcated lesions with a largest diameter ≥1.5 cm, or
* 1 clearly demarcated lesion with a largest diameter ≥2.0 cm
* The patient was not previously treated for indolent lymphoma (with the exception of a single course of local radiation therapy not exceeding 2 adjacent lymph node regions).
* The patient has adequate hematologic and hepatic function.
* The patient has Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* The patient has serum creatinine of 2.0 mg/dL or less or creatinine clearance of 30 mL/min or more, based on the Cockcroft-Gault method, or from a 24-hour urine collection.
* The patient is willing to comply with contraception requirements.

Key Exclusion Criteria:

The patient:

* Has small lymphocytic lymphoma or mantle cell lymphoma.
* Has documented history of central nervous system (CNS) lymphomatous involvement.
* Has or has had an active malignancy, other than NHL, within the past 3 years except for localized prostate cancer without evidence of bone metastases, bladder, cervical, or breast carcinoma in-situ, or non-melanoma skin cancer .
* Has New York Heart Association (NYHC) Class III or IV heart failure, uncontrolled arrythmias or unstable angina, electrocardiographic evidence of active ischemia or active conduction system abnormalities, or myocardial infarction within the last 6 months.
* Has known human immunodeficiency virus (HIV) infection.
* Has acute or chronic hepatitis B or hepatitis C infection.
* Is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* Has any serious uncontrolled, medical or psychological disorder that would impair the ability of the subject to receive study drugs.
* Has received another investigational agent within 30 days of study entry.
* Has known hypersensitivity to mannitol.
* Has Ann Arbor stage I disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon
Locations (38):
- United States (34):
  - Birmingham Hematology and Oncology Associates, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Hematology Oncology, P.C., Stamford, Connecticut
  - University Cancer Institute, Boynton Beach, Florida
  - Florida Cancer Institute - New Hope, New Port Richey, Florida
  - Dublin Hematology Oncology Care P.C., Dublin, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - Georgia Cancer Specialists, Tucker, Georgia
  - Cancer Care and Hematology Specialists of Chicagoland, Niles, Illinois
  - Siouxland Hematology-Oncology Assoc. LLP, Sioux City, Iowa
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Carroll County Cancer Center, Westminster, Maryland
  - Columbia Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Somerset Hematology Oncology Associates, Somerville, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center, Lake Success, New York
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pittsburgh Medical Center - Cancer Institute, Pittsburgh, Pennsylvania
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Longview Cancer Center, Longview, Texas
  - Joe Arrington Cancer Research, Lubbock, Texas
  - Texas Oncology, P.A., McAllen, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Oncology, Waco, Texas
  - Texas Oncology, P.A., Webster, Texas
  - US Oncology Research - Texoma Cancer Center, Wichita Falls, Texas
  - Fairfax/Northern Virginia Hematology/Oncology, Fairfax, Virginia
  - Yakima Valley Memorial Hospital/North Start Lodge, Yakima, Washington
- Belgium (2):
  - Cephalon Investigational Site, Brussels
  - Cephalon Investigational Site, Ghent
- Israel (2):
  - Cephalon Investigational Site, Haifa
  - Cephalon Investigational Site, Nahariya

REFERENCES:
- [Derived] Czuczman MS, Kahanic S, Forero A, Davis G, Munteanu M, Van Den Neste E, Offner F, Bron D, Quick D, Fowler N. Results of a phase II study of bendamustine and ofatumumab in untreated indolent B cell non-Hodgkin's lymphoma. Ann Hematol. 2015 Apr;94(4):633-41. doi: 10.1007/s00277-014-2269-8. Epub 2015 Jan 30. PMID 25630297

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bendamustine and Ofatumumab
Started | 50
Safety Set (Enrolled and Treated) | 49
Completed | 45
Not Completed | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bendamustine and Ofatumumab
Number analyzed (Participants) | 49
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.77)
Age, Customized [Number; unit: participants]
  <65 years | 31
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 45
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Pacific Islander | 0
  Black | 2
  White | 44
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR), as Determined by the International Working Group (IWG) Criteria As Assessed by Investigators
Description: The IWG criteria (Cheson et al 2007) for a CR is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A PR is at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase should be observed in the size of other nodes, liver or spleen, and no new sites of disease should be observed.
Time Frame: up to Week 32
Population: Safety population of participants who were treated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine and Ofatumumab
Number analyzed (Participants) | 49
percentage of participants | 90 [77.8 to 96.6]

2. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), as Determined by the International Working Group (IWG) Criteria As Assessed by Investigators
Description: The IWG criteria (Cheson et al 2007) for a CR is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: up to Week 32
Population: Safety population of participants who were treated
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bendamustine and Ofatumumab
Number analyzed (Participants) | 49
percentage of participants | 67 [52.6 to 80.1]

ADVERSE EVENTS:
Time Frame: up to 39 weeks
Arm/Group | Bendamustine and Ofatumumab
Serious Adverse Events (participants affected / at risk) | 14/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine and Ofatumumab (N=49)
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Diplopia (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Faeces discoloured (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Infusion related reaction (General disorders) | 2
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Device dislocation (General disorders) | 1
Fatigue (General disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 1
Bacterial sepsis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Oxygen saturation decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hot flush (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bendamustine and Ofatumumab (N=49)
Neutropenia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 7
Anaemia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Lymphopenia (Blood and lymphatic system disorders) | 3
Tachycardia (Cardiac disorders) | 5
Palpitations (Cardiac disorders) | 3
Eye irritation (Eye disorders) | 4
Nausea (Gastrointestinal disorders) | 29
Constipation (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 12
Vomiting (Gastrointestinal disorders) | 12
Abdominal pain (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4
Stomatitis (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 26
Infusion related reaction (General disorders) | 20
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 6
Chills (General disorders) | 6
Asthenia (General disorders) | 4
Drug hypersensitivity (Immune system disorders) | 5
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 4
White blood cell count decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 7
Weight decreased (Investigations) | 4
Haemoglobin decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 12
Dizziness (Nervous system disorders) | 10
Dysgeusia (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 7
Anxiety (Psychiatric disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8
Urticaria (Skin and subcutaneous tissue disorders) | 8
Periorbital oedema (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 5
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.